CLINICAL TRIAL: NCT01121900
Title: A Randomized, Two-way Crossover Study to Compare the Bioavailability of 300 mg Trazodone Hydrochloride Extended-release Caplets (Containing Contramid®) (Administered as a Single Dose) and 100 mg Trazodone Hydrochloride Immediate-release Tablets (Administered Three Times Daily) Under Fasting Conditions
Brief Title: A Study to Compare the Bioavailability of 300 mg Trazodone Hydrochloride Extended-release Caplets and 100 mg Trazodone Hydrochloride Immediate-release Tablets (Administered Three Times Daily)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04ACL1-010
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — Trazodone

ARMS (2):
- Trazodone HCl OAD (Experimental): OAD: Once A Day
  Interventions: Drug: Trazodone HCl
- Trazodone HCl (Apotex Corp.) (Active Comparator)
  Interventions: Drug: Trazodone HCl

INTERVENTIONS:
Drug: Trazodone HCl — Dosage form: Extended-release caplets containing 300 mg trazodone HCl
  Dose: 300 mg trazodone HCl extended-release caplets (one caplet) at 23:30 on Day 1 of the test product treatment period following a fasting period of at least 4 hours.
  Other Names: Oleptro
  Arms: Trazodone HCl OAD
Drug: Trazodone HCl — Dosage form: Immediate-release tablets containing 100 mg trazodone HCl
  Dose: 100 mg trazodone HCl immediate-release tablets (one tablet per dosing time) at 23:30 on Day 1, at 07:30 and 15:30 on Day 2 of the reference product treatment period.
  Arms: Trazodone HCl (Apotex Corp.)

SUMMARY:
The objective of this study was to compare the pharmacokinetic profiles of the test product, 300 mg trazodone hydrochloride (HCl) extended-release caplets (containing Contramid®), when administered as a single dose, and the reference product, 100 mg trazodone HCl immediate-release tablets (Apotex Corp), when administered three times daily. For this purpose the rate and extent of absorption of trazodone and formation of m-chlorophenylpiperazine (mCPP) after administration of the two formulations, were compared under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18 to < 56 years of age.
* Body mass within 10% of the ideal mass in relation to height and age, according to Body Mass Index.
* Body mass not less than 53 kg.
* Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the laboratory reference ranges for the relevant laboratory tests (unless the investigator considered the deviation to be irrelevant for the purpose of the study).
* Normal 12-lead electrocardiogram (ECG) and vital signs, or abnormalities, which the investigator did not consider a disqualification for participation in the study.
* Willingness to undergo a pre- and post-study physical examination and laboratory investigations.
* Ability to comprehend and willingness to sign both statements of informed consent (for screening and period-related procedures).
* Non-smoker or past smoker who stopped the use of any form of tobacco, including snuff or similar products, at least 3 months before entering the study.
* For females, the following conditions had to be met:

  1. Had been surgically sterilized or undergone a hysterectomy, or
  2. Was of childbearing potential, and all of the following conditions were met:

     1. Had a negative pregnancy test at screening. If this test was positive, the subject was to be excluded from the study before receiving study medication. In the rare circumstance that a pregnancy was discovered after the subjects received the study medication, every attempt was to be made to follow such subjects to term.
     2. Had to agree to use an accepted method of contraception (i.e., spermicide and barrier methods or spermicide and non-hormonal intrauterine contraceptive device). The subject had to agree to continue with the same method throughout the study. Hormonal contraceptives were not allowed.
  3. Females not of childbearing potential could also have been included if they had no menstrual period for one year and were considered as post-menopausal.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to have limited the validity of consent to participate in the study or to have limited the ability to comply with protocol requirements.
* History of, or current compulsive alcohol abuse (> 10 drinks weekly), or regular exposure to other substances of abuse.
* Use of any medication, prescribed or over-the-counter, within 2 weeks prior to the first administration of study medication except if this would not have affected the outcome of the study in the opinion of the investigator. Hormonal contraceptive agents were not allowed.
* Participation in another study with an experimental drug, where the last administration (of previous study medication) was within 8 weeks before the first administration of study medication.
* Treatment within the previous 3 months with any drug with a well-defined potential for adversely affecting a major organ or system.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity to the study medication or any related medication.
* History of bronchial asthma.
* History of epilepsy.
* History of porphyria.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to have influenced the study outcome.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of study medication.
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
* Positive testing for HIV and/or Hepatitis B and/or Hepatitis C.
* Positive urine screen for drugs of abuse.
* Positive urine screen for tobacco use.
* A serum pregnancy test (beta human chorionic gonadotropin [β-HCG]) either positive or not performed or lactation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

REFERENCES:
- See also: Approved Labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=17925

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Trazodone Contramid® OAD) First: Trazodone Contramid® OAD (Once-A-Day) test product (300 mg tablet once daily) dosed in first treatment phase followed by Trazodone IR (Apotex Corp.) reference product (100 mg tablet thrice daily) dosed in the second treatment phase. A drug-free period of 7 to 14 calendar days separated the last administration of study medication in treatment period 1 and the first administration of study medication in treatment period 2.
  IR = Immediate Release.
- Reference (Trazodone IR [Apotex Corp.]) First: Trazodone IR (Apotex Corp.) reference product (100 mg tablet thrice daily) dosed in first treatment phase followed by Trazodone Contramid® OAD (Once-A-Day) test product (300 mg tablet once daily) dosed in the second treatment phase. A drug-free period of 7 to 14 calendar days separated the last administration of study medication in treatment period 1 and the first administration of study medication in treatment period 2.
  IR = Immediate Release.
Period: First Intervention Period
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR [Apotex Corp.]) First
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Washout Period of 7 Days
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR [Apotex Corp.]) First
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention Period
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR [Apotex Corp.]) First
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Test first and Reference first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.2 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Region of Enrollment [Number; unit: participants]
  South Africa | 26

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence Based Cmax
Description: Cmax = Maximum plasma concentration. Measured in nanogram per milliliter (ng/mL).
Time Frame: 68 hours
Population: The dataset for pharmacokinetic analysis comprised the 23 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Trazodone Contramid® OAD: Trazodone Contramid® OAD test product (300 mg tablet administered once daily) dosed in either first intervention period or second intervention period. A drug-free period of 7 to 14 calendar days separated the last administration of study medication in Phase 1 and the first administration of study medication in Phase 2.
- Trazodone IR (Apotex Corp.): Trazodone IR (Apotex Corp.) reference product (100 mg tablet administered thrice daily)dosed in either first intervention period or second intervention period. A drug-free period of 7 to 14 calendar days separated the last administration of study medication in Phase 1 and the first administration of study medication in Phase 2.
Arm/Group | Trazodone Contramid® OAD | Trazodone IR (Apotex Corp.)
Number analyzed (Participants) | 23 | 23
ng/mL | 1230.7 (499.1) | 2947.7 (734.7)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD vs Trazodone IR (Apotex Corp.); Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LSmeans) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter Cmax is between 80% and 125%; Mean ratio = 39.8, 90% CI 2-sided [34.4 to 46.0] — Test/reference (%)

2. Primary Outcome: Bioequivalence Based on AUC(0-tlast)
Description: AUC(0-tlast) = Area under the plasma concentration curve (AUC) vs (versus) time data pairs, where tlast is the time of the last quantifiable concentration.
  Measured in nanogram x hours per milliliter (ng*h/mL).
Time Frame: 68 hours
Population: The dataset for pharmacokinetic analysis comprised the 23 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Trazodone Contramid® OAD | Trazodone IR (Apotex Corp.)
Number analyzed (Participants) | 23 | 23
hr*ng/mL | 28138.4 (8400.0) | 34272.4 (9792.8)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD vs Trazodone IR (Apotex Corp.); Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LSmeans) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter AUC(0-tlast) is between 80% and 125%; Mean ratio = 80.9, 90% CI 2-sided [74.2 to 88.3] — Test/reference (%)

3. Primary Outcome: Bioequivalence Based on AUC(0-∞)
Description: AUC(0-∞) = Area under the plasma concentration curve vs time data pairs, with extrapolation to infinity (∞).
  Measured in nanogram x hours per milliliter (ng*h/mL).
Time Frame: 68 hours
Population: The dataset for pharmacokinetic analysis comprised the 23 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Trazodone Contramid® OAD | Trazodone IR (Apotex Corp.)
Number analyzed (Participants) | 23 | 23
h*ng/mL | 29672.5 (8373.8) | 35258.5 (10067.4)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD vs Trazodone IR (Apotex Corp.); Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LSmeans) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter AUC(0-∞) is between 80% and 125%; Mean ratio = 83.5, 90% CI 2-sided [76.5 to 91.1] — Test/reference (%)

4. Secondary Outcome: Area Under the Plasma Concentration vs. Time Data Pairs, for the First 24 Hours [AUC(0-24)]
Time Frame: 24 hours
Population: The dataset for pharmacokinetic analysis comprised the 23 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Trazodone Contramid® OAD | Trazodone IR (Apotex Corp.)
Number analyzed (Participants) | 23 | 23
h*ng/mL | 18331.0 (4966.4) | 24602.2 (6097.5)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Time Frame: 68 hours
Population: The dataset for pharmacokinetic analysis comprised the 23 subjects who completed the study as per protocol.
Measure: Median (Full Range); unit: Hours
Arm/Group | Trazodone Contramid® OAD | Trazodone IR (Apotex Corp.)
Number analyzed (Participants) | 23 | 23
Hours | 9.00 (3.64) [2.00 to 16.02] | 8.33 (1.66) [8.33 to 16.33]

6. Secondary Outcome: Apparent Terminal Elimination Rate Constant (λz)
Description: The elimination rate constant of trazodone (Lamda z). It is the ratio of clearance to volume of distribution and is expressed in units of 1/hour. This constant is used in half-life calculations.
Time Frame: 68 hours
Population: The dataset for pharmacokinetic analysis comprised the 23 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Trazodone Contramid® OAD | Trazodone IR (Apotex Corp.)
Number analyzed (Participants) | 23 | 23
1/hour | 0.064 (0.018) | 0.090 (0.024)

7. Secondary Outcome: Apparent Terminal Half-life (t½.z)
Description: The elimination half-life (T½z) of trazodone in plasma (time it takes for the concentration of trazodone to fall to half), expressed in hours.
Time Frame: 68 hours
Population: The dataset for pharmacokinetic analysis comprised the 23 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Trazodone Contramid® OAD | Trazodone IR (Apotex Corp.)
Number analyzed (Participants) | 23 | 23
Hours | 11.8 (3.7) | 8.3 (2.5)

ADVERSE EVENTS:
Description: A total of 24 subjects were exposed to Trazodone Contramid® OAD during the study (13 during first intervention period and 11 during second intervention period).
  A total of 25 subjects were exposed to Trazodone IR (Apotex Corp.) during the study (13 during first intervention period and 12 during second intervention period).
Arm/Group | Trazodone Contramid® OAD | Trazodone IR (Apotex Corp.)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 7/24 | 8/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trazodone Contramid® OAD (N=24) | Trazodone IR (Apotex Corp.) (N=25)
Dizziness (Nervous system disorders) | 5 (6) | 4 (5)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication based on the results of this study is envisaged, approval from the Sponsor will be obtained and a draft manuscript will be submitted to the sponsor for scrutiny and comment. The choice of scientific journal will be mutually agreed on by the principal investigator and the sponsor.